CLINICAL TRIAL: NCT04461483
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dose and Multiple Doses With Titration of TAK-935 in Healthy Japanese Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dose and Multiple Doses With Titration of TAK-935 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-1004; U1111-1252-8555 (Other: WHO); JapicCTI-205349 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1, Cohort 1; TAK-935 200 mg (Experimental): Part 1, Cohort 1; TAK-935 200 mg, tablets, orally once on Days 1 in fasted state.
  Interventions: Drug: TAK-935
- Part 1, Cohort 2; TAK-935 600 mg (Experimental): Part 1, Cohort 2; TAK-935 600 mg, tablets, orally once on Days 1 in fasted state.
  Interventions: Drug: TAK-935
- Part 1, Cohort 3; TAK-935 1200 mg (Experimental): Part 1, Cohort 3; TAK-935 1200 mg, tablets, orally once on Days 1 in fasted state.
  Interventions: Drug: TAK-935
- Part 1, Cohort 1-3; Placebo (Placebo Comparator): Part 1, Cohort 1-3; TAK-935 placebo-matching tablets, orally once on Days 1 in fasted state.
  Interventions: Drug: Placebo
- Part 2, Cohort 4: TAK-935 100 mg (Experimental): Part 2, Cohort 4: TAK-935 100 mg, tablets, orally twice on Days 1-7 in fasted state with multiple doses with titration.
  Interventions: Drug: TAK-935
- Part 2, Cohort 4: TAK-935 200 mg (Experimental): Part 2, Cohort 4: TAK-935 200 mg, tablets, orally twice on Days 8-14 in fasted state with multiple doses with titration.
  Interventions: Drug: TAK-935
- Part 2, Cohort 4: TAK-935 300 mg (Experimental): Part 2, Cohort 4: TAK-935 300 mg, tablets, orally twice on Days 15-21 in fasted state with multiple doses with titration.
  Interventions: Drug: TAK-935
- Part 2, Cohort 4: Placebo (Placebo Comparator): Part 2, Cohort 4: TAK-935 placebo-matching tablets, orally twice on Days 1-21 in fasted state.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-935 — TAK-935 Tablets
  Arms: Part 1, Cohort 1; TAK-935 200 mg; Part 1, Cohort 2; TAK-935 600 mg; Part 1, Cohort 3; TAK-935 1200 mg; Part 2, Cohort 4: TAK-935 100 mg; Part 2, Cohort 4: TAK-935 200 mg; Part 2, Cohort 4: TAK-935 300 mg
Drug: Placebo — TAK-935 placebo-matching tablets
  Arms: Part 1, Cohort 1-3; Placebo; Part 2, Cohort 4: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TAK-935 with single ascending doses (Part 1) and multiple doses with titration (Part 2).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935 tablet. TAK-935 tablet is being tested in Japanese healthy adult men. This study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TAK-935 with single ascending doses (Part 1) and multiple doses with titration (Part 2).

The study will enroll up to 33 participants in total (Part 1 + 2). In Part 1, participants will be randomly assigned (by chance, like flipping a coin) to one of these treatment cohorts/groups;

* Cohort 1: Single dose of TAK-935 at 200 mg or placebo (fasted)
* Cohort 2: Single dose of TAK-935 at 600 mg or placebo (fasted)
* Cohort 3: Single dose of TAK-935 at 1200 mg or placebo (fasted)

In Part 2, participants will be randomly assigned to one of these treatment groups;

- Cohort 4: Multiple doses with titration of TAK-935 or placebo at 100 mg twice daily (BID) from Day 1 to Day 7, 200 mg BID from Day 8 to Day 14 and 300 mg BID from Day 15 to Day 21 (fasted).

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 36 days for Part 1 and 63 days for Part 2. Participants will be hospitalized for 5 days in Part 1 and 26 days in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must understand the study procedures and agree to participate by providing written informed consent.
2. The participant must be willing and able to comply with all study procedures and restrictions.
3. The participant must be a Japanese healthy adult male or female, aged 20 to 55 years, inclusive, at the time of informed consent.
4. The participant must have a body mass index (BMI) >=18.5 and =<25.0 kg/m^2 at the Screening Visit.
5. The participant must be a current nonsmoker who has not used tobacco- or nicotine-containing products (eg, nicotine patch) for at least 6 months prior to the first dose of study drug or first invasive procedure.
6. The participant must be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead electrocardiogram, and vital sign measurements performed at the Screening Visit and prior to the first dose of study drug.
7. The participant must meet the following birth control requirements:

   * Is a male participant who is sterile or agrees to use an appropriate method of contraception, including a condom with spermicidal cream or jelly, from the first dose of study drug until 90 days after the last dose of study drug. No restrictions are required for a vasectomized male participant provided the participant is at least 1-year postbilateral vasectomy procedure prior to the first dose of study drug. A male participant whose vasectomy procedure was performed less than 1 year prior to the first dose of study drug must follow the same restrictions as a nonvasectomized man. Appropriate documentation of surgical procedure should be provided.
   * Is a male participant who agrees to not donate sperm from the first dose of study drug until 90 days after the last dose of study drug.
   * Is a female participant of nonchildbearing potential, defined by at least 1 of the following criteria:

     1. Postmenopausal (defined as 12 months of spontaneous amenorrhea in females aged >45 years or >=6 months of spontaneous amenorrhea in females aged >45 years with serum follicle-stimulating hormone [FSH] levels >40 mIU/mL). Appropriate documentation of follicle-stimulating hormone levels should be required.
     2. Hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
     3. Had a tubal ligation with appropriate documentation of surgical procedure.
     4. Congenital conditions such as uterine aplasia etc.

Exclusion Criteria:

1. Has a history of clinically significant endocrine, gastrointestinal (including motility disorder and intestinal obstruction), cardiovascular (including arrhythmia), hematological, hepatic, immunological, renal, respiratory, genitourinary, major neurological (including stroke, epileptic seizure), or degenerative ophthalmological abnormalities or diseases
2. Has participated in another investigational trial within 4 weeks or 5 half-lives (whichever is longer) before the pretrial visit (Screening). The 4-week or 5 half-lives window will be derived from the date of the last trial procedure and/or AE related to the trial procedure in the previous trial to the pretrial/Screening Visit of the current trial.
3. Is an employee or immediate family member (eg, spouse, parent, child, sibling) of the sponsor.
4. Has a history of cancer (malignancy).
5. Has any lifetime history of a suicide attempt, or have suicidal ideation or, any suicidal behavior within 12 months, or who are at significant risk to commit suicide, as judged by the investigator using the Columbia Suicide Severity Rating Scale (C-SSRS) or is clinically judged by the investigator to be at risk for suicide.
6. Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
7. Has a positive alcohol or drug screen.
8. Had major surgery, donated or lost whole blood prior to the start of study drug administration as any of below:

   For both male and female participants, >=200 mL within 4 weeks (28 days) For male participants, >=400 mL within 12 weeks (84 days), >=800 mL in total within 52 weeks (364 days) For female participants, >=400 mL within 16 weeks (112 days). >=400 mL in total within 52 weeks (364 days)
9. Had gastrointestinal surgery that could impact the absorption of study drug.
10. Has a history of a major psychiatric disorder as diagnosed utilizing Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria.
11. Has a known hypersensitivity to any component of the formulation of TAK-935 or related compounds.
12. Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies, beginning approximately 7 days before administration of the initial dose of study drug, throughout the trial (including washout intervals between trial periods), until the Follow-up Visit.
13. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
14. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
15. Has a substance abuse disorder.
16. Has a QTcF >450 msec confirmed with one repeat testing, at the Screening Visit.
17. Had abnormal Screening or Day -1 laboratory values that suggested a clinically significant underlying disease or participant with the following laboratory abnormalities: ALT and/or AST >1.5 time ULN.
18. Has tested positive for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, HIV antibody/antigen, or serologic reactions for syphilis at Screening.
19. In the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 13 August 2020 to 14 November 2020.
Pre-assignment Details: Healthy Japanese participants were enrolled in the study into two parts: Single Ascending Dose (SAD) (Part 1) and Multiple Dose (MD) titration (Part 2) to receive TAK-935 tablets or TAK-935 placebo-matching tablets.
Groups:
- Part 1, SAD, Cohorts 1 to 3: Placebo: TAK-935 placebo-matching tablet, orally, once on Day 1 in fasted state.
- Part 1, SAD, Cohort 1: TAK-935 200 mg: TAK-935 200 milligram (mg), tablet, orally, once on Day 1 in fasted state.
- Part 1, SAD, Cohort 2: TAK-935 600 mg: TAK-935 600 mg, tablet, orally, once on Day 1 in fasted state.
- Part 1, SAD, Cohort 3: TAK-935 1200 mg: TAK-935 1200 mg, tablet, orally, once on Day 1 in fasted state.
- Part 2, MD, Cohort 4: Placebo: TAK-935 placebo-matching tablets, orally, twice daily on Days 1 to 21 in fasted state.
- Part 2, MD, Cohort 4: TAK-935: TAK-935 100 mg, tablets, orally, twice daily on Days 1 to 7, then up-titrated to TAK-935 200 mg, tablets, orally, twice daily, on Days 8 to 14, further up-titrated to TAK-935 300 mg, tablets, orally, twice daily on Days 15 to 21 as multiple doses with titration in the fasted state.
Period: Part 1 (Day 1)
Arm/Group | Part 1, SAD, Cohorts 1 to 3: Placebo | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg | Part 2, MD, Cohort 4: Placebo | Part 2, MD, Cohort 4: TAK-935
Started | 6 | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Day 1 to 21)
Arm/Group | Part 1, SAD, Cohorts 1 to 3: Placebo | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg | Part 2, MD, Cohort 4: Placebo | Part 2, MD, Cohort 4: TAK-935
Started | 0 | 0 | 0 | 0 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Part 1, SAD, Cohort 1: TAK-935 200 mg: TAK-935 200 mg, tablet, orally, once on Day 1 in fasted state.
- Total: Total of all reporting groups
Arm/Group | Part 1, SAD, Cohorts 1 to 3: Placebo | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg | Part 2, MD, Cohort 4: Placebo | Part 2, MD, Cohort 4: TAK-935 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 6 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.43) | 39.0 (12.71) | 31.5 (14.11) | 41.5 (11.20) | 37.7 (8.39) | 33.5 (7.48) | 37.1 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 3 | 6 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 6 | 6 | 3 | 6 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 3 | 6 | 33
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.5 (6.95) | 169.8 (4.02) | 167.0 (8.39) | 173.3 (5.61) | 173.7 (1.53) | 168.2 (2.64) | 170.1 (5.74)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 63.78 (4.392) | 59.88 (4.212) | 58.75 (5.410) | 65.47 (7.750) | 65.70 (1.778) | 61.38 (2.865) | 62.2 (5.311)
Body-mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.98 (1.755) | 20.77 (1.206) | 21.05 (0.822) | 21.75 (1.473) | 21.77 (0.306) | 21.75 (1.571) | 21.49 (1.326)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 5 | 3 | 6 | 4 | 3 | 4 | 25
  Former Smoker | 1 | 3 | 0 | 2 | 0 | 2 | 8
Alcohol Classification [Count of Participants; unit: Participants]
  Had Daily Consumption | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Had a Few Times Per Week | 0 | 1 | 1 | 2 | 0 | 2 | 6
  Had a Few Times Per Month | 4 | 2 | 3 | 2 | 0 | 1 | 12
  Had no Consumption | 2 | 3 | 2 | 0 | 3 | 3 | 13
Caffeine Classification [Count of Participants; unit: Participants]
  Had Caffeine | 2 | 3 | 0 | 3 | 1 | 1 | 10
  Had no Caffeine | 4 | 3 | 6 | 3 | 2 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Part 1: Baseline up to Day 8; Part 2: Baseline up to Day 35
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Part 2, MD, Cohort 4: TAK-935 100 mg: TAK-935 100 mg, tablets, orally, twice daily on Days 1 to 7 in fasted state.
- Part 2, MD, Cohort 4: TAK-935 200 mg: TAK-935 200 mg, tablets, orally, twice daily on Days 8 to 14 in fasted state following TAK-935 100 mg, tablet, orally, twice daily.
- Part 2, MD, Cohort 4: TAK-935 300 mg: TAK-935 300 mg, tablets, orally, twice daily on Days 15 to 21 in fasted state following TAK-935 200 mg, tablet, orally, twice daily.
Arm/Group | Part 1, SAD, Cohorts 1 to 3: Placebo | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg | Part 2, MD, Cohort 4: Placebo | Part 2, MD, Cohort 4: TAK-935 100 mg | Part 2, MD, Cohort 4: TAK-935 200 mg | Part 2, MD, Cohort 4: TAK-935 300 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 33.33 | 16.7 | 33.33

2. Secondary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug and had at least 1 estimable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg
Number analyzed (Participants) | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 413.2 (202.4) | 3001 (47.3) | 9278 (48.1)

3. Secondary Outcome: Part 2, Cmax: Maximum Observed Plasma Concentration for TAK-935
Time Frame: Days 7, 14, and 21 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: The PK analysis set included all participants who received at least 1 dose of study drug and had at least 1 estimable PK parameter. As planned data for this outcome measure was collected, analyzed and reported for dose level TAK-935-100 mg on Day 7, dose level TAK-935-200 mg on Day 14, and TAK-935-300 mg on Day 21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2, MD, Cohort 4: TAK-935 100 mg | Part 2, MD, Cohort 4: TAK-935 200 mg | Part 2, MD, Cohort 4: TAK-935 300 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 146.5 (113.1) | 835.5 (73.8) | 1945 (37.7)

4. Secondary Outcome: Part 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK analysis set included all participants who received at least 1 dose of study drug and had at least 1 estimable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg
Number analyzed (Participants) | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL) | 512.7 (100.8) | 3538 (45.8) | 10590 (42.1)

5. Secondary Outcome: Part 1, AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Infinity for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 539.2 (97.2) | 3603 (45.1) | 10660 (42.0)

6. Secondary Outcome: Part 1, AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 517.8 (99.4) | 3538 (45.8) | 10540 (41.0)

7. Secondary Outcome: Part 2, AUCtau,ss: Area Under the Plasma Concentration-time Curve During the Dosing Interval at Steady State for TAK-935
Time Frame: Days 7, 14, and 21 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2, MD, Cohort 4: TAK-935 100 mg | Part 2, MD, Cohort 4: TAK-935 200 mg | Part 2, MD, Cohort 4: TAK-935 300 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 202.3 (54.6) | 788.6 (48.9) | 1960 (27.7)

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after the first dose of study drug (Baseline) up to Day 8 in Part 1, and up to Day 35 in Part 2
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part 1, SAD, Cohort 1-3: Placebo: TAK-935 placebo-matching tablet, orally, once on Day 1 in fasted state.
- Part 2, MD, Cohort 4: Placebo: TAK-935 placebo-matching tablets, orally, twice daily on Days 1to 21 in fasted state.
Arm/Group | Part 1, SAD, Cohort 1-3: Placebo | Part 1, SAD, Cohort 1: TAK-935 200 mg | Part 1, SAD, Cohort 2: TAK-935 600 mg | Part 1, SAD, Cohort 3: TAK-935 1200 mg | Part 2, MD, Cohort 4: Placebo | Part 2, MD, Cohort 4: TAK-935 100 mg | Part 2, MD, Cohort 4: TAK-935 200 mg | Part 2, MD, Cohort 4: TAK-935 300 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 2/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, SAD, Cohort 1-3: Placebo (N=6) | Part 1, SAD, Cohort 1: TAK-935 200 mg (N=6) | Part 1, SAD, Cohort 2: TAK-935 600 mg (N=6) | Part 1, SAD, Cohort 3: TAK-935 1200 mg (N=6) | Part 2, MD, Cohort 4: Placebo (N=3) | Part 2, MD, Cohort 4: TAK-935 100 mg (N=6) | Part 2, MD, Cohort 4: TAK-935 200 mg (N=6) | Part 2, MD, Cohort 4: TAK-935 300 mg (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04461483/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04461483/SAP_001.pdf